CLINICAL TRIAL: NCT02281799
Title: Thiopurine Induced Pancreatitis in IBD Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No Participants Enrolled
Sponsor: Shaare Zedek Medical Center (Other)
Collaborators: Sydney Children's Hospitals Network (Other); Christchurch Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Thiopurine_Pancreatitis
Record Dates: First submitted 2014-10-23; First posted 2014-11-04 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2017-10

CONDITIONS: Pancreatitis; Inflammatory Bowel Diseases
Keywords: Azathioprine (AZA); 6-mercaptopurine (6-MP); Thiopurine-S-methyltransferase (TPMT); Xanthine oxidase (XO); 6-thioguanine (6-TGN); 6-methyl-mercaptopurine (6-MMP); inflammatory bowel disease (IBD); acute pancreatitis (AP); inosine triphosphate pyrophosphohydrolase (ITPA); rheumatoid arthritis (RA); systemic lupus erythematosis (SLE); Crohn's disease (CD); ulcerative colitis (UC)
MeSH Terms: conditions — Pancreatitis; Inflammatory Bowel Diseases; Arthritis, Rheumatoid; Crohn Disease; Colitis, Ulcerative | interventions — Azathioprine; Mercaptopurine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label (Experimental): 10 patients diagnosed with IBD, treated previously with thiopurines and ceased treatment due to suspected thiopurine-induced pancreatitis.
  Patients will be commenced on an alternative thiopurine to that used initially,. The medications will be commenced at standard dose (ie Azathioprine 2.5mg/kg/day, 6-MP 1.5mg/kg/day).
  Interventions: Drug: Azathioprine

INTERVENTIONS:
Drug: Azathioprine — Patients will be commenced on an alternative thiopurine to that used initially, according to the standard dosing schedule used by their IBD clinician.
  For example, if the initial thiopurine-related pancreatitis occurred while taking Azathioprine, the patient will be restarted on 6-MP, and vice versa.
  Other Names: 6-mercaptopurine

SUMMARY:
Azathioprine (AZA) and its metabolite 6-mercaptopurine (6-MP) were developed over 50 years ago by Gertrude Elion and George Hitchings and were initially used clinically in the management of childhood leukemia and organ transplantation.

The first case report of 6-MP use in inflammatory bowel disease (IBD) was from 1962 , and since then the use of thiopurines has been well established in the management of moderate to severe IBD.

Thiopurines offer an inexpensive and effective treatment option for maintenance of remission of IBD in comparison to biological agents which may be 30 times more expensive .

Although 50-60% of IBD patients respond to thiopurines, a significant proportion of patients will not tolerate them due to various adverse effects . The adverse effects of thiopurines may be dose related, patient related or idiosyncratic.

The immunosuppressive effects of thiopurines also increase the rates of opportunistic infections.

Thiopurines are also associated with a higher rate of malignancies, particularly a malignant Burkitt-like lymphoma, related to Epstein-Barr virus infection . Other adverse effects of thiopurine relate to allergic phenomenon.

An idiosyncratic adverse effect of thiopurine use is acute pancreatitis (AP).

Acute inflammation of the pancreas defined by INSPPIRE criteria:

requiring 2 of:

1. Abdominal pain compatible with AP
2. Serum amylase and/or lipase ≥ 3 times upper limits of normal
3. Imaging findings of AP

Drug induced AP is the assumed diagnosis when no other cause of AP can be found, the patient is taking a drug known to be associated with AP, and symptoms resolve after drug discontinuation. If pancreatitis re-occurs on re-exposure, the drug is definitely considered the cause.

While drugs are considered a rare cause of AP and most cases are mild and self limited , there is an 8 fold higher risk of AP in IBD patients treated with AZA . Thiopurine induced AP is usually detected within 4 weeks of starting treatment.

However in the case of thiopurine induced AP, there has been no clear understanding of the mechanism.

Thiopurine induced AP is generally considered an indication to cease thiopurine therapy, due to the assumed risk of recurrence of AP on reintroduction.

There exists several case reports and anecdotal evidence that reintroducing thiopurines following an assumed thiopurine associated AP can be well tolerated.

The investigators hypothesize that AZA and/or 6-MP can be safely reintroduced in the management of IBD patients following thiopurine-induced pancreatitis.

If in the past the patients were treated with AZA, they will now be commenced on 6-MP, and if in the past they were treated with 6-MP, they will be commenced on AZA.

DETAILED DESCRIPTION:
The research protocol extends for up to 3.5 months, during which the participant will attend 5 clinic visits at Shaare Zedek Medical Centre: screening visit, week 0, week 4, week 8 and week 12.

During the screening visit, all patients identified who meet the exclusion and inclusion criteria and who agree to participate in the study, will have their medical records reviewed for previous clinical or biochemical evidence of pancreatitis, both related, and unrelated to thiopurine use.

Patients will undergo a physical examination, baseline blood tests including measurement of lipase and/or amylase, liver biochemistry and fasting lipid profile. If not already tested, the patients TPMT activity will be tested. Participants will also have a baseline abdominal ultrasound to confirm normal anatomy and absence of cholelithiasis At week 0, if there are no clinical, biochemicals or ultrasound suggestions of pancreatitis, the participant will be commenced on an alternative thiopurine from what was used in the past. That is, if in the past they were treated with AZA, they will now be commenced on 6-MP, and if in the past they were treated with 6MP, they will be commenced on AZA. The medications will be commenced at standard dose (ie AZA 2.5mg/kg/day, 6MP 1.5mg/kg/day). Depending on the specific situation, and assuming all relevant information is available, the screening visit may be merged with the week 0 visit.

In weeks 1, 2, 3 and 6 will have blood tests (full blood count and liver biochemistry) performed at a local clinic, and the investigator will be in telephone contact with the participant to discuss the results and to discuss if there are any adverse effects of the medication.

In weeks 4, 8 and 12 the participant will attend clinic with the investigator for a medical history, clinical examination and review of blood tests (blood count and liver enzymes).

In the event of any new onset upper abdominal pain or emesis, patients will be instructed to present to their nearest medical facility for blood tests (including serum amylase and/or lipase) and an ultrasound, if clinically indicated, to contact the investigator and to consider cessation of the thiopurine.

At the end of the 3 month period, if patients show no sign of pancreatitis, they will revert to regular monitoring of thiopurine therapy as per their treating gastroenterologist.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with IBD, treated previously with thiopurines, and ceased treatment due to suspected thiopurine-induced pancreatitis
* Ability to consent to and participate in the study and follow study procedures
* Age 5-60 years

Exclusion Criteria:

* Previous severe pancreatitis requiring prolonged hospital admission or intensive care involvement, or Ranson's criteria ≥ 3
* No clinical need to reintroduce a thiopurine for management of IBD at the time of the study (e.g. stable on another medication, or mild phenotype of disease), based on clinical assessment of treating gastroenterologist
* Diagnosis of recurrent pancreatitis syndrome
* Diabetes mellitus or any other neuropathy which may dampen the clinical presentation of pancreatitis
* Known or suspected allergy or intolerance to thiopurines, besides previous pancreatitis
* Any other laboratory or clinical condition that the investigator considers clinically significant that could impact the outcome of the study or the safety of the patient.

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Number of participants demonstrating biochemical or clinical evidence of pancreatitis | 3 month period following intervention

SECONDARY OUTCOMES:
Number of participants with adverse events or hospitalization experienced as a result of intervention | 3 month period following intervention

CONTACTS AND LOCATIONS:
Overall Officials: Oren Ledder, MD, Principal Investigator — Shaare Zedek
Locations (1):
- Shaare Zedek, Jerusalem, Israel